CLINICAL TRIAL: NCT06440993
Title: The CLEAN-DUCT / TRITICC-3 Trial - Phase IIa, Prospective, Single Arm, Open Label, Non-randomized, Multi-center Pilot Study of Durvalumab (MEDI4736) + Intraductal Radiofrequency Ablation (ID-RFA) in Extrahepatic Cholangiocarcinoma
Brief Title: Durvalumab + Intraductal Radiofrequency Ablation (ID-RFA) in Extrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Universitätsklinikum Düsseldorf, Germany (Unknown); Universitätsklinikum Köln (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEAN-DUCT / TRITICC-3; 2023-509165-21-00 (EU CTIS Number); ESR-23-22156 (Other Grant/Funding Number: AstraZeneca); IKF-t070 (Other: IKF Trial ID)
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Extrahepatic Cholangiocarcinoma; Unresectable Perihilar or Ductal CCA
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Gemcitabine; Cisplatin; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- systemic plus ID-RFA (Experimental): systemic treatment: - combination treatment for 8 cycles (Q3W):
  * Gemcitabine, 1,000 mg/m2 IV, on day 1 and 8,
  * Cisplatin, 25 mg/m2 IV, on day 1 and 8
  * Durvalumab, 1,500 mg IV, on day 1 followed by
  * Durvalumab maintenance, 1,500 mg IV, PLUS • 2 endoscopic intraductal RFA
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Durvalumab; Procedure: ID-RFA

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine, 1,000 mg/m2 IV
Drug: Cisplatin — Cisplatin, 25 mg/m2 IV
Drug: Durvalumab — Durvalumab, 1,500 mg IV
Procedure: ID-RFA — endoscopic intraductal RFA

SUMMARY:
The present clinical trial is a prospective, investigator-initiated, single-arm, open-label, multicenter phase II trial. Patients with unresectable perihilar and/or ductal CCA with indication for bile duct stenting and palliative systemic therapy as determined by the local multidisciplinary team (MDT), who already resolved cholestasis due to RFA + Stent will be enrolled.

We hypothesize that in patients with extrahepatic cholangiocarcinoma, the use of a combination radiofrequency ablation followed by systemic treatment with chemotherapy plus durvalumab might further increase the anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

1. Patient* has given written informed consent.
2. Patient is ≥ 18 years of age at time of signing the written informed consent.
3. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
4. Patient has been diagnosed with histologically or cytologically confirmed

   1. histologically or cytologically confirmed cholangiocarcinoma as adenocarcinoma of pancreatobiliary type
   2. unresectable perihilar and/or ductal cholangiocarcinoma with indication for bile duct stenting and palliative systemic therapy as determined by the local multidisciplinary team (MDT) and already resolved cholestasis due to RFA + stent
5. Patient tolerated RFA prior to inclusion and is eligible for repeat RFA during the study (does not have any contraindications) as determined by investigator.
6. Patient is eligible for palliative systemic therapy based on clinical and laboratory parameters (except hyperbilirubinemia) as determined by the local MDT
7. Patient has a ECOG ≤ 1.
8. Patient has life expectancy of ≥ 12 weeks
9. Patient has body weight > 30 kg
10. Adequate blood count, liver-enzymes, and renal function:

    1. ANC > 1,500 cells/μL without the use of hematopoietic growth factors
    2. Platelet count ≥ 100 x 109/L (>100,000 per mm3)
    3. Hemoglobin ≥ 9 g/dL
    4. Serum total bilirubin ≤ 3x upper normal limit (ULN) (biliary drainage is allowed for biliary obstruction; elevated bilirubin should be caused by obstruction not impaired liver function as assessed by albumin and INR values)
    5. Albumin levels ≥ 2.8 g/dL
    6. Patients not receiving therapeutic anticoagulation must have an INR< 2.0 ULN and PTT < 1.5 ULN within 7 days prior to randomization. The use of full dose anticoagulants is allowed as long as the INR or PTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least three weeks at the time of inclusion
    7. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional ULN unless liver metastases are present, in which case it must be ≤ 5x ULN
    8. Serum Creatinine ≤ 1.5 x ULN and a calculated creatinine clearance rate ≥ 60 mL /min
11. Female patients defined as women of childbearing potential (WOCBP) or male patients with WOCBP partners must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 6 months after the last dose of chemotherapy or for at least 3 months after last dose of durvalumab, whatever happens last. Male patients must refrain from donating sperm during this same period. Male patients with a pregnant partner must agree to remain abstinent or to use a condom for the duration of the pregnancy.

Exclusion Criteria:

1. Patient received previous or simultaneous endobiliary treatment other than RFA (e.g. PDT or brachytherapy)
2. Patient received previous systemic therapy with a PD-1, PD-L1 inhibitor (including durvalumab) or CTLA4 inhibitor or classical chemotherapy agents like platinum, fluoropyrimidine or gemcitabine-based regimens.
3. Patient receives any concurrent chemotherapy, investigational product or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer related conditions (e.g., hormone replace therapy) is acceptable.
4. Patient has known hypersensitivity to any component of the durvalumab formulation as well as a known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion protein and/or any known contraindication (including hypersensitivity) to gemcitabine or cisplatin.
5. Patient has history of primary immunodeficiency
6. Patient has stage B cirrhosis according to Child-Pugh criteria (or worse) or cirrhosis (of any grade) with a history of hepatic encephalopathy or clinically significant ascites resulting from cirrhosis. Clinically significant ascites is defined as ascites resulting from cirrhosis requiring diuretics or paracentesis.
7. Patient has any unresolved NCI CTCAE grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and laboratory values defined in the inclusion criteria

   1. Patients with grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the Lead Investigator
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Lead Investigator.
8. Patient had a prior allogeneic bone marrow transplantation or prior solid organ transplantation.
9. Patient has active or history of autoimmune or inflammatory disorders (including, but not limited to, inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis]) . The following are exceptions:

   1. Patients with vitiligo or alopecia
   2. Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement
   3. Patients with any chronic skin condition that does not require systemic therapy
   4. Patients with celiac disease controlled by diet alone
   5. Patients without active disease in the last 5 years may be included but only after consultation with the Lead Investigator
10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | at 12 months
  Overall survival rate after 12 months (OS@12months) defined as proportion of patients alive 12 months after enrollment

SECONDARY OUTCOMES:
Progression-free survival (PFS) | at study end
  Progression-free survival (PFS) defined as time from enrollment to the date of disease progression or death from any cause
Overall survival (OS) | at study end
  Overall survival (OS) Defined as time from enrollment to the date of death from any cause
Incidence and nature of adverse events using NCI CTCAE 5.0 | through study completion, up to 3years
  Assessment of safety of the treatment as determined by the incidence, nature, causality, frequency, timing and severity of adverse events using NCI CTCAE 5.0
Time to cholangitis | from enrollment to first cholangitis event, up to 3 years
  Time to cholangitis Defined as time from enrollment to the date of confirmed cholangitis
To assess quality of life (QoL) data from patients using EORTC QLQ-BIL21 | through study completion, up to 3years
  To assess quality of life (QoL) data from patients using EORTC QLQ-BIL21
To assess quality of life (QoL) data from patients using EORTC QLQ-C30 | through study completion, up to 3years
  To assess quality of life (QoL) data from patients using EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin SE Al-Batran, Prof. Dr., Study Chair — Frankfurter Institut fuer Klinische Krebsforschung IKF GmbH
Locations (10):
- Germany (10):
  - Uniklinik RWTH Aachen, Aachen
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Krankenhaus Nordwest, Frankfurt
  - Universitätsmedizin Göttingen, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - UKSH Campus Lübeck, Lübeck
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Universitätsklinik Münster, Münster

IPD SHARING:
Plan to Share IPD: No